CLINICAL TRIAL: NCT00652548
Title: Utility of Bedside Ultrasound to Diagnose Clavicle Fractures in the Pediatric Emergency Department
Brief Title: Use of Ultrasound to Evaluate Clavicle Fractures in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Keith Cross, Assistant Professor, University of Louisville
Other Study IDs: 08-0007; IRB #08-0007; NHRO #1310
Record Dates: First submitted 2008-03-28; First posted 2008-04-03 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Fractures
Keywords: Clavicle; Fracture; Ultrasound; Radiation
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This studies investigates the hypothesis that bedside ultrasound is as accurate as plain x-rays for diagnosing clavicle fractures in children in a pediatric emergency department. Children with shoulder injuries are enrolled and receive both an ultrasound imaging (experimental) and x-rays (standard-of-care) to see if ultrasound has the same (or better)accuracy, with less cost, time, and radiation.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-18 years
* Pain from recent shoulder/clavicle injury
* Intact neurovascular exam
* Radiographs performed as part of normal ED evaluation

Exclusion Criteria:

* Hemodynamic instability
* Multisystem trauma
* Altered mental status
* Open wounds to injured shoulder
* Developmental delay
* Prior radiographs at another clinic/hospital for this injury
* Previous clavicle fracture on the affected side
* Ultrasound gel allergy
* Non-English-speaking parents/child (unable to give informed consent)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children age 1-18 years presenting to a tertiary center pediatric emergency department complaining of recent traumatic shoulder injury.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Comparison of a blinded reviewer's interpretation of bedside US images to an attending radiologist's interpretation of radiographs | Single visit to emergency department

SECONDARY OUTCOMES:
Unblinded real-time bedside US by the ED physician vs. radiographs | Single ED visit
Interoperator reliability between the blinded reviewer and bedside ED physician | Single ED visit
FACES pain score for pain for US vs. radiographs for children ≥ 5 yrs | Single ED visit

CONTACTS AND LOCATIONS:
Overall Officials: Keith P Cross, MD, Principal Investigator — University of Louisville
Locations (1):
- Kosair Children's Hospital, Louisville, Kentucky, United States